CLINICAL TRIAL: NCT04800861
Title: Glycemic Control in Diabetic Hospitalized Patients: a Cross Sectional Study
Brief Title: Glycemic Control in Diabetic Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: AlFayhaa General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1121
Record Dates: First submitted 2021-03-05; First posted 2021-03-16 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Diabetes Mellitus
Keywords: diabetes mellitus; hyperglycemia; glycemic control; inpatient
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the advanced management of diabetes and new innovative anti-hyperglycemic therapy hyperglycemia remains a culprit factor affecting the outcome of patients admitted to the hospital in general wards. Efforts from health care providers to assess and control blood sugar by a simplified method such as certified point of care hand-sized glucometers is the fruitful protocol if the results near the target that is endorsed by well-known diabetes societies. In non-critically patients the premeal blood sugar ≤140 mg /dl and ≤ 180 mg /dl after a meal. The unstable economy and political crises with the pandemic of Covid-19 making us use a glucometer to monitor and control the fluctuation of blood sugar in order to decrease the burden on the patients and health care providers in the form of a stay in the hospital and minimize wasting laboratory resources.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the hospital

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: diabetic patients admitted in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
glycemic control | From hospital admission to hospital discharge for a median of 7 days and up to 1 month
  percentage of patients with glucose measurement (Random Blood Sugar, RBS, Fasting Blood Sugar, FBS) between 140-180 measured with bedside glucometers preferably before meals and at 6 am for fasting blood sugars or as directed by the physician

SECONDARY OUTCOMES:
average blood glucose value per ward | From hospital admission to hospital discharge for a median of 7 days and up to 1 month
  average blood glucose value per ward (medical vs. surgical vs ICU/CCU
average per patient | From hospital admission to hospital discharge for a median of 7 days and up to 1 month
  average blood glucose levels per patient

CONTACTS AND LOCATIONS:
Overall Officials: AbdulSattar J Yousif, MD, Study Chair — Al-Fayhaa teaching hospital; Ali Hussein A Alhamza, MD, Study Chair — Al-Fayhaa teaching hospital
Locations (1):
- AlFayhaa Teaching hospital, Basra, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
unidentified patient data will be shared if requested